CLINICAL TRIAL: NCT00739128
Title: Intradermal Immunization Against Hepatitis B Virus in Celiac Disease- a Randomized Controlled Trial
Brief Title: Response to Hepatitis B Vaccine in Celiac Disease Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Believed that a better study was to compare the response to engerix B vs Sci-B-Vac vaccine in this patient group.
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Ari Silbermintz, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15363.ct.il
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Celiac Disease
Keywords: celiac disease; hepatitis B vaccine
MeSH Terms: conditions — Celiac Disease; Hepatitis B | interventions — Hepatitis B Vaccines; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): celiac patients who did not respond to initial hepatitis B vaccine series , will receive repeat hep B vaccine via intramuscular route
  Interventions: Biological: hepatitis B vaccine (EngerixB)
- 2 (Active Comparator): celiac patients who did not respond to initial hepatitis B vaccine series , will receive repeat hep B vaccine via intradermal route
  Interventions: Biological: hepatitis B vaccine (EngerixB)

INTERVENTIONS:
Biological: hepatitis B vaccine (EngerixB) — A dose of 10mcg (0.5 ml) of the recombinant HBV vaccine will be administered intramuscular at zero, one and six months intervals
  Other Names: EngerixB, GSK
  Arms: 1
Biological: hepatitis B vaccine (EngerixB) — A dose of 10mcg (0.5 ml) of the recombinant HBV vaccine will be administered intradermally in the deltoid region at zero, one and six months intervals
  Other Names: (EngerixB, GSK)
  Arms: 2

SUMMARY:
Celiac disease and infection with hepatitis B virus (HBV) are very prevalent worldwide and carry a high morbidity rate. It has been recently shown that patients with celiac disease very often fail to develop immunity after standard vaccination for HBV during infancy. In this study, we will evaluate whether a second vaccination series via a different route of administration (into the skin rather than the muscle) results in a better immunological response in celiac patients. Eligible patients will be randomized to receive a 3-dose vaccination series into the skin or to the muscle. Rate of responders and level of immunity will be compared. This study will facilitate better protection of celiac patients to this potentially deadly virus.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 1 year of age with confirmed diagnosis of celiac disease by characteristic symptoms, serology and small bowel biopsy.
* Completion of the IM HBV vaccine series in infancy.
* HBsAb titer of ≤10mIU/mL at the time of enrollment.

Exclusion Criteria:

* Immunocompromised subjects or those receiving medications that may modulate or suppress the immune system (i.e. azathiopurine, 6-MP, steroids).
* Inability to obtain written informed consent and patients' assent, as appropriate by the maturity age.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
1. The primary endpoint of the study will be comparison of the geometric mean titers of anti-HBs between the intradermal and the intramuscular groups. | two years

SECONDARY OUTCOMES:
1. Rate of responders four weeks after the completion of the series 2. Rate and characteristics of adverse drug reactions 3. Numerical increase in the antibodies titer before and after vaccination 4. Rate of responders in the cross over phase | two years

CONTACTS AND LOCATIONS:
Overall Officials: Maskit Bar Meir, MD, Principal Investigator — Shaheed Ziaur Rahman Medical College; Ari Silbermintz, Principal Investigator — Shaheed Ziaur Rahman Medical College
Locations (1):
- SZMC, Jerusalem, Israel